CLINICAL TRIAL: NCT06799975
Title: Effects of a Single Session of Physiotherapy on Pain, Disability and Psychological Risk Factors in Patients Operated for Lumbar Spondylolisthesis: a Randomized Controlled Study
Brief Title: Effects of a Single Session of Physiotherapy on Patients Operated for Lumbar Spondylolisthesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF23/00
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Spondylolisthesis
Keywords: lumbar spondylolisthesis; physiotherapy; disability; psychological factors; randomized controlled trial
MeSH Terms: conditions — Spondylolisthesis | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor was unaware of the participant's intervention group, as was the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education (Experimental): The intervention consists of a single physiotherapy session before discharge.
  Interventions: Other: Education
- Usual care (Active Comparator): Usual discharge procedures
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Education — Patients in the "education" group will have a meeting with a physiotherapist at the end of the T1 evaluation, which will take place in a suitable room that ensures privacy is maintained. During this meeting, the physiotherapist will provide the patient with advice regarding their return home and will suggest simple exercises to activate/maintain the abdominal and lower back muscles, to be performed at home until the next visit, one month after the surgery. These exercises are part of standard clinical practice and should be routinely performed by patients who undergo lumbar spinal fusion in the period following the surgery. Additionally, the patient will have the opportunity to communicate, via email or phone, with the physiotherapist until the follow-up appointment with the spine surgeon (scheduled for one month later).
  Arms: Education
Other: Usual Care — The usual discharge procedures consist of a brief interview with the neurosurgeon during which instructions are provided on how to manage the first month after the surgery.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to investigate whether a meeting with physiotherapist before hospital discharge can improve the post-operative outcomes in patients who have undergone lumbar fusion surgery for spondylolisthesis.

The main question it aims to answer is:

* The primary endpoint investigated is the degree of disability measured using the ODI-I one month after the surgical intervention.
* The secondary endpoints are the level of pain measured using the NRS scale at 1 and 3 months post-surgery; disability at 3 months measured using the ODI-I questionnaire; physical function assessed using the UWT at 1 and 3 months post-surgery; psychological factors such as self-efficacy and fear of movement measured using the TSK and PSEQ-I at 1 and 3 months after lumbar fusion surgery; health status and quality of life measured at 3 months with the HADS-I and SF-36-I questionnaires; and the patient's satisfaction regarding their hospital stay, assessed using a PREMs questionnaire administered at the time of discharge.

The "usual care" group will instead be discharged by the spinal surgeon following the standard procedures.

The physiotherapist will provide the patient with advice regarding their return home and will suggest simple exercise to be performed at home until the next visit, one month after surgery. Additionally, the patient will have the opportunity to communicate, either by email or phone, with the physiotherapist until the follow-up visit with the spinal surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients who have undergone lumbar fusion surgery due to monosegmental lumbar spondylolisthesis.

Exclusion Criteria:

* Patients who have undergone previous lumbar surgeries
* Patients operated on for other lumbar pathologies
* Patients with pre-existing neurological deficits not related to the condition being treated
* Patients with systemic conditions (inflammatory, infectious, neoplastic, etc.) or neuromuscular disorders
* Patients with cognitive deficits or psychiatric disorders
* Patients who do not speak Italian fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Oswestry Disability Index | From enrollment to the 1 month follow-up
  Validated questionnaire to assess the patient's disability

SECONDARY OUTCOMES:
Changes in Numeric Rating Scale | From enrollment to the 1 month follow-up
  Scale assessing the perceived pain
Changes in Numeric Rating Scale | From enrollment to the 3 months follow-up
  Scale assessing the perceived pain
Changes in Numeric Rating Scale | From 1 month to the 3 months follow-up
  Scale assessing the perceived pain
Changes in Oswestry Disability Index | From enrollment to the 3 months follow-up
  Validated questionnaire to assess the patient's disability
Changes in Oswestry Disability Index | From 1 month follow-up to the 3 months follow-up
  Validated questionnaire to assess the patient's disability
Changes in Hospital Anxiety and Depression Scale | From enrollment to the 1 month follow-up
  Validated questionnaire to assess the anxiety and depression
Changes in Hospital Anxiety and Depression Scale | From enrollment to the 3 months follow-up
  Validated questionnaire to assess the anxiety and depression
Changes in Hospital Anxiety and Depression Scale | From 1 month follow-up to the 3 months follow-up
  Validated questionnaire to assess the anxiety and depression
Changes in Pain Self-Efficacy Questionnaire | From enrollment to the 1 month follow-up
  Validated questionnaire to assess the self-efficacy
Changes in Pain Self-Efficacy Questionnaire | From enrollment to the 3 months follow-up
  Validated questionnaire to assess the self-efficacy
Changes in Pain Self-Efficay Questionnaire | From 1 month follow-up to the 3 months follow-up
  Validated questionnaire to assess the self-efficacy
Changes in Short Form Health Survey 36 | From enrollment to the 3 months follow-up
  Validated questionnaire to assess the quality of life
Changes in Tampa Scale of Kinesiophobia | From enrollment to the 1 month follow-up
  Validated questionnaire to assess the kinesiophobia
Changes in Tampa Scale of Kinesiophobia | From enrollment to the 3 months follow-up
  Validated questionnaire to assess the kinesiophobia
Changes in Tampa Scale of Kinesiophobia | From 1 month follow-up to the 3 months follow-up
  Validated questionnaire to assess the kinesiophobia
Changes in Up and Walking Test | From enrollment to the 1 month follow-up
  Physical test to assess the patient's functional status. The test consists of standing up from a chair without using the upper limbs, walking 5 meters, turning around, walking back, and sitting down again without using the upper limbs.
Changes in Up and Walking Test | From enrollment to the 3 months follow-up
  Physical test to assess the patient's functional status. The test consists of standing up from a chair without using the upper limbs, walking 5 meters, turning around, walking back, and sitting down again without using the upper limbs.
Changes in Up and Walking Test | From 1 month follow-up to the 3 months follow-up
  Physical test to assess the patient's functional status. The test consists of standing up from a chair without using the upper limbs, walking 5 meters, turning around, walking back, and sitting down again without using the upper limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy